CLINICAL TRIAL: NCT02750566
Title: Comparing the Effect of Osteopathic Manipulative Medicine (OMM) Versus Counseling in the Treatment of Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Sheldon Yao, Associate Profession, Chair of the Department of Osteopathic Manipulative Medicine, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1139
Record Dates: First submitted 2015-12-04; First posted 2016-04-25 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Post-Concussion Symptoms; Distorted; Balance
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Manipulation, Osteopathic; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): A board certified NMM/OMM or FP/OMM physician will perform an osteopathic structural exam and osteopathic treatment for a 30 minute session. The investigators will follow a generalized protocol for diagnosis and treatment of the head, neck, spine, rib cage, and pelvis. The following techniques will be included in the treatment protocol, OA (Occipitoatlantal) decompression, V-Spread, venous sinus drainage, balanced membranous tension (BMT), cranial lifts, CV4, and a mix of balanced ligamentous tension (BLT), muscle energy techniques, facilitated positional release, articulatory techniques (ART), high-velocity low-amplitude, and counterstrain to address any somatic dysfunctions.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Counseling (Active Comparator): For the control group, an investigator will complete a 30-minute counseling session with the subject. The focus of discussion will be from the CDC's "What to expect after a concussion" article. Other resources that will also be used come from the American Academy of Family Physicians (AAFP), FamilyDoctor.org, and the Brain Care Center. Each counseling session will follow the same protocol. The counseling session will provide subject with similar face-to-face time with the OMT arm.
  Interventions: Other: Counseling

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Manual treatment of musculoskeletal restrictions that may be prevent proper healing post-concussion.
  Other Names: Osteopathic Manipulative Medicine
  Arms: Osteopathic Manipulative Treatment
Other: Counseling — Patients will be counseled on concussion awareness, symptoms, and treatment for 30 minutes by a physician.
  Arms: Counseling

SUMMARY:
Concussion or mild traumatic brain injury (TBI) is a challenging injury for physicians to manage and is among the most serious disabling neurological disorders. Physician awareness regarding manifestations of TBI and subsequent treatment are paramount to reduce the burden of disease. Advancements in treatment of mild TBI have been slow with a lack of consensus on treatment methods that show universal success. This gap in treatment choices provides an opportunity for osteopathic manipulative treatment (OMT) to fill. OMT is a hands-on manual therapy that can be integrated to help treat post-concussive symptoms. Previous studies have shown that OMT can help resolve imbalance and tinnitus in elderly populations and case studies have shown that this manual therapy may assist in patient recovery. The investigators hypothesize that OMT will decrease return to play/work time, will show an improvement in balance, and will decrease concussion symptoms as compared to counseling.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to investigate the effectiveness of osteopathic manipulative treatment (OMT) in improving concussion-related symptoms.

Previous studies and case reports have found a positive effect of OMT on resolving concussion-like symptoms such as vertigo, imbalance, and tinnitus. It is hypothesized that OMT improves proprioceptive input from the cervical spine and joints and sensory input from the internal auditory meatus. The investigators propose to further investigate this relationship in order to quantify the effect of OMT through the SMART Balance Master and return to play/work time. As this is a pilot study, the investigators intend to determine if a correlation exists between OMT and return to work/play and SMART Balance Master scores.

Specifically, the investigators have three main aims for this study:

Specific Aim #1: OMT will show a statistically significant improvement balance as measured by the SMART Balance Master scores pre- and post-OMT

Specific Aim #2: OMT will decrease concussion symptom as measured by surveys

Specific Aim #3: OMT will decrease return to play/work time in concussed subjects compared to standard.

Background/Rationale:

Concussion or mild traumatic brain injury (TBI) is a challenging injury for physicians to manage. It is undetectable by traditional imaging techniques, and there are limited treatment options. A concussion results from a biomechanical force directed towards the head that precedes and contributes to neurologic dysfunction, including impairment in the level of consciousness. However, a loss of consciousness is not a requirement for the diagnosis.

The CDC estimates the annual burden of concussion in the United States to be roughly 1.4-3.8 million. Over the past decade, the CDC also reports a 70% increase in TBI emergency department visits, as well as an increase in TBI-related hospitalizations. Other studies have determined the prevalence of individuals with chronic concussion problems in the US is 5.3 million. Importantly, these figures should be considered an underestimate as patients with milder injuries often do not seek treatment.

The mechanism of concussion involves a primary and secondary phase of tissue injury. A primary injury is immediate and irreversible, resulting from acceleration/deceleration mechanical damage. Secondary injuries result from non-mechanical damage derived from neuronal cell membrane disruption and axonal stretch. The membrane defects result from secondary injury and lead to ionic influx and accumulation of toxic substances such as glutamate within the nervous system. Individuals with mild concussion recover within a few days; however, 15% of patients with mild concussion suffer from long-term complications largely due to the secondary phase of injury.

Recent literature has studied the role of restricted cerebral blood flow and inflammation on perpetuating the symptoms of a concussion. Meier et al. discovered an inverse relationship between cerebral blood flow in the dorsal midinsular cortex and the time to return to play. Other studies have investigated the role of inflammation, through the production of reactive oxygen species, that not only contribute to the initial injury but also potentiate its own pathological course. These studies highlight potential mechanisms that could be targeted to decrease symptoms and improve outcomes.

Treatment for mild concussion in the past has been limited to bed rest. Previous studies have noted that bed rest following a concussion does not improve recovery time and, if continued for too long, can negatively impact recovery. Some pilot projects have reported promising findings such as decreased 30-day mortality with progesterone. Through a meta-analysis of non-surgical interventions following a mild TBI, Nygren-de Boussard et al. found that there are poor randomized controlled trials or comparison groups to indicate any intervention can provide therapeutic benefit. Furthermore, evidence supports a more individualized approach when treating post-concussive symptoms.

Alternative or complementary treatments encompass a variety of individual approaches for different patients including herbal supplements, homeopathy, hyperbaric oxygen, arts and recreational therapies, meditation practice, and Tai Chi Chuan. Empirical literature on alternative treatments for mild concussion is sparse, with many studies either insufficiently powered or poorly controlled. The widespread use and popularity of these treatment options and their potential to help treat concussions demands further scientific investigation.

Osteopathic manipulative treatment (OMT) is defined in the Glossary of Osteopathic Terminology as "the therapeutic application of manually guided forces by an osteopathic physician to improve physiologic function and/or support homeostasis that has been altered by somatic dysfunction." Somatic dysfunctions, or restrictions of skeletal or myofascial structures, disrupt the normal function of vascular, lymphatic and neural components related to or that pass through these structures. By treating somatic dysfunctions, OMT aims to remove musculoskeletal (MSK) restrictions which allow for increased blood flow and lymphatic drainage and decreased nerve impingements. Somatic dysfunctions in the cranium and spine can contribute to patient's concussion symptoms including dizziness and tinnitus. Treatment of somatic dysfunctions with OMT, targeting structures involved with concussion-related symptoms, may be another treatment option that can be offered to these patients.

Evidence has supported the use of the SMART Balance Master as a validated tool to measure balance. Fraix et al. used the SMART Balance Master by NeuroCom® to quantify the beneficial effect of OMT on improving patients' balance and dizziness. The SMART Balance Master® can be used to quantify changes in balance before and after OMT. The Sensory Organization Test (SOT) is one assessment tool that can measure three different aspects of balance and posture: somatosensory, visual, and vestibular. The complete protocol for SOT can be found on the NeuroCom® website.

The ImPACT test is a widely used tool to help detect and assess the severity of concussion in athletes. This computerized test is administered to athletes routinely to establish a baseline of memory and cognitive function, and administered again in the suspicion of a concussion in order to evaluate the difference in cognitive function. The test is widely used and has been shown to be an effect adjunct test for evaluation of concussion as part of a comprehensive medical diagnosis involving other testing methods.

The SCAT-3 (sport concussion assessment tool - 3rd edition) is an improved version of a widely used aid for physicians for evaluating concussion severity and progress. The test is a combination of patient-reported symptom evaluation as well as an objective cognitive and physical exam.

The King-Devick Test objectively measures visual tracking and saccadic eye movements (rapid movement of the eye between fixation points). The test was originally developed in 1976 by eye care specialists to help evaluate reading disabilities as they related to oculomotor movement. Since 2011, the test has been used as a rapid sideline screening tool for concussion in a variety of sports, based on the findings that concussion is associated with many neuro-ophthalmologic signs. Many studies have shown the King-Devick Test to be a valid aid in detecting and evaluating concussions.

It is with these tools, the investigators aim to measure the effects of OMT on post-concussion symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years age
* Subject has suffered from non-life threatening head trauma head trauma resulting in current concussion-related symptoms
* Subject is evaluated and diagnosed with a concussion
* Subject has been cleared to participate in the study by the physician/neurologist having excluded any potential emergent conditions

Exclusion Criteria:

* The subject has no absolute contraindications to osteopathic manipulative treatment, such as skull fracture, cervical fracture, signs of intracranial bleeding, cervical dissection, or stroke
* The subject suffered from any of the following at the time of event leading to concussion:

  * Loss of consciousness >2 minutes in the field
  * Seizures
  * Intractable vomiting
  * Paralysis
* The subject has been diagnosed with an underlying neurodegenerative condition that may confound test results (e.g.. Parkinson's Disease, Alzheimer's Disease)
* The subject has a current or previous spinal cord injury
* The subject is unable to complete the assessment tools
* The subject is pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
SMART Balance Master balance scores pre and post intervention arm | change from the pre-intervention score after the intervention, measured at each visit through study completion, an average of 1 week after the initial visit
  OMT should show a statistically significant improvement in balance as measured by SMART Balance Master balance scores as measured by change pre and post procedure

SECONDARY OUTCOMES:
Post-concussion symptoms as measured by ImPACT | measured on day 1, day 3, and day 7 post concussion
  OMT should decrease concussion symptoms as measured by subject responses on this performance test as measured by change pre and post procedure
Post-concussion symptoms as measured by King-Devick | measured on day 1, day 3, and day 7 post concussion
  OMT should decrease concussion symptoms as measured by subject responses on this performance test as measured by change pre and post procedure.
Post-concussion symptoms as measured by SCAT-3 | measured on day 1, day 3, and day 7 post concussion
  OMT should decrease concussion symptoms as measured by subject responses on this survey as measured by change pre and post procedure.

OTHER OUTCOMES:
Return to play time | Up to 90 days
  Players will be tracked for eventual clearance to return to play and OMT should decrease return to play time.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Yao, DO, Principal Investigator — NYITCOM
Locations (1):
- Academic Helath Care Center - Sports Medicine Center, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fraix M, Gordon A, Graham V, Hurwitz E, Seffinger MA. Use of the SMART Balance Master to quantify the effects of osteopathic manipulative treatment in patients with dizziness. J Am Osteopath Assoc. 2013 May;113(5):394-403. PMID 23667193
- [Background] King D, Gissane C, Hume PA, Flaws M. The King-Devick test was useful in management of concussion in amateur rugby union and rugby league in New Zealand. J Neurol Sci. 2015 Apr 15;351(1-2):58-64. doi: 10.1016/j.jns.2015.02.035. Epub 2015 Feb 26. PMID 25748294
- [Background] Schatz P, Pardini JE, Lovell MR, Collins MW, Podell K. Sensitivity and specificity of the ImPACT Test Battery for concussion in athletes. Arch Clin Neuropsychol. 2006 Jan;21(1):91-9. doi: 10.1016/j.acn.2005.08.001. Epub 2005 Sep 6. PMID 16143492
- [Background] Guskiewicz KM, Register-Mihalik J, McCrory P, McCrea M, Johnston K, Makdissi M, Dvorak J, Davis G, Meeuwisse W. Evidence-based approach to revising the SCAT2: introducing the SCAT3. Br J Sports Med. 2013 Apr;47(5):289-93. doi: 10.1136/bjsports-2013-092225. PMID 23479486
- [Background] Corps KN, Roth TL, McGavern DB. Inflammation and neuroprotection in traumatic brain injury. JAMA Neurol. 2015 Mar;72(3):355-62. doi: 10.1001/jamaneurol.2014.3558. PMID 25599342
- [Derived] Mazzeo S, Silverberg C, Oommen T, Moya D, Angelo N, Zwibel H, Mancini J, Leder A, Yao SC. Effects of Osteopathic Manipulative Treatment on Sleep Quality in Student Athletes After Concussion: A Pilot Study. J Am Osteopath Assoc. 2020 Aug 11. doi: 10.7556/jaoa.2020.100. Online ahead of print. PMID 32780797
- [Derived] Yao SC, Zwibel H, Angelo N, Leder A, Mancini J. Effectiveness of Osteopathic Manipulative Medicine vs Concussion Education in Treating Student Athletes With Acute Concussion Symptoms. J Am Osteopath Assoc. 2020 Aug 7. doi: 10.7556/jaoa.2020.099. Online ahead of print. PMID 32766808